CLINICAL TRIAL: NCT00430781
Title: A Phase II, Open-Label, Randomized, Multicenter Trial of Pazopanib (GW786034) in Combination With Lapatinib (GW572016) Compared to Pazopanib Monotherapy and Lapatinib Monotherapy in Subjects With FIGO Stage IVB or Recurrent or Persistent Cervical Cancer With Zero or One Prior Chemotherapy Regimen
Brief Title: Pazopanib Plus Lapatinib Compared to Lapatinib Alone and Pazopanib Alone In Subjects With Metastatic Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEG105281
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Results first posted 2011-03-14 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Neoplasms, Uterine Cervix; Metastatic Cervical Cancer
Keywords: pazopanib; ErB1/ErB2; lapatinib; persistent; VEGF; recurrent; metastatic cervical cancer; advanced; FIGO Stage IVB
MeSH Terms: conditions — Neoplasms; Uterine Cervical Neoplasms; Recurrence | interventions — pazopanib; Lapatinib

ARMS (3):
- Combination arm (Experimental): Pazopanib plus lapatinib
  Interventions: Drug: lapatinib (GW572016)
- Lapatinib monotherapy (Active Comparator): Lapatinib
  Interventions: Drug: lapatinib (GW572016)
- Pazopanib monotherapy (Active Comparator): Pazopanib
  Interventions: Drug: pazopanib (GW786034)

INTERVENTIONS:
Drug: pazopanib (GW786034)
  Arms: Pazopanib monotherapy
Drug: lapatinib (GW572016)
  Arms: Combination arm; Lapatinib monotherapy

SUMMARY:
This study is being conducted to compare the efficacy and safety of pazopanib in combination with lapatinib with that of lapatinib alone or pazopanib alone in subjects with metastatic cervical cancer

DETAILED DESCRIPTION:
A Phase II, Open-Label, Randomized, Multicenter Trial of Pazopanib (GW786034) in Combination with Lapatinib (GW572016) Compared to Pazopanib Monotherapy and Lapatinib Monotherapy in Subjects with International Federation of Gynecology (FIGO) Stage IVB or Recurrent or Persistent Cervical Cancer with Zero or One Prior Chemotherapy Regimen for Advanced/Recurrent Disease

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria are met:
* Signed, written informed consent prior to performing any study-related procedures
* Female subjects ≥18 years of age
* FIGO Stage IVB, or recurrent or persistent cervical cancer
* Life expectancy of at least 12 weeks
* ECOG status of 0 or 1.
* Histologically confirmed FIGO Stage IVB, or recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥ 20 mm when measured by conventional techniques, including palpitation, plain x-ray, CT and MRI, or ≥10 mm when measured by spiral CT.
* At least one "target lesion" to be used to assess response as defined by Response Evaluation Criteria in Solid Tumors (RECIST; Terasse, 2000). Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
* Received 0 or 1 prior chemotherapy regimen for metastatic disease.
* Note: Chemotherapy given in combination with radiation therapy as a radiosensitizer does not count toward this prior therapy limit
* Recovered from the effects of surgery or chemotherapy. At least three weeks must have elapsed from the last administration of chemotherapy.
* Adequate organ and bone marrow function as defined in Table 1.
* Table 1:(Definitions for Adequate Organ Function)
* System:(Laboratory Values)
* Hematologic: Absolute neutrophil count (ANC)(≥ 1.5 X 109/L)Hemoglobin1(≥9 g/dL)Platelets(≥100 X 109/L)
* Hepatic: Total bilirubin (≤1.5 X ULN)AST and ALT (≤2.5 X ULN)
* Renal: Calculated creatinine clearance2 (≥50 mL/min)
* Urine protein3 (Negative, trace or +1 by dipstick urinalysis or <1.0 gram determined by 24 hour urine protein analysis.)
* Subjects may not have had a transfusion within 7 days of screening assessment.
* Calculated by Cockcroft Gault formula See Appendix 7: Renal Function Tests
* A patient should first be screened with dipstick urinalysis. If urine protein by dipstick analysis is ≥2+, then a 24-hour urine protein must be assessed and 24 hour urine protein must be <1 g protein to be eligible.
* Ability to swallow and retain oral medication.
* A female is eligible to enter and participate in this study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:
* A hysterectomy
* A bilateral oophorectomy (ovariectomy)
* A bilateral tubal ligation
* Is post-menopausal (total cessation of menses for ≥ 1 year)
* Childbearing potential, has a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:
* An intrauterine device with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigation product, through the dosing period, and for at least 21 days after the last dose of investigational product.
* Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

Note: Oral contraceptives are not reliable due to potential drug-drug interactions.

* Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow-up as outlined in the protocol. Procedures conducted as apart of routine clinical management of the patient (e.g., blood count, imaging study) and obtained prior to signed informed consent may be utilized for screening purposes provided these tests are obtained as specified in the protocol

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Neuroendocrine or small cell carcinoma of the cervix.
* Prior use of any biologic therapy with VEGF, VEGFR, or ErbB1/ErbB2 inhibitors.
* Concurrent cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, and tumor embolization).
* Concurrent treatment with an investigational agent or participation in another clinical trial.
* Use of an investigational anti-cancer drug within 28 days or 5 half-lives, whichever is longer, preceding the first dose of study medication.
* Has taken or is taking prohibited medications listed in the protocol.
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with patient's safety, obtaining informed consent or compliance to the study.
* History of another malignancy. Note: Patients who have had another malignancy and have been disease-free for 5 years, or patients with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis. Routine screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated.
* Malabsorption Syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
* Active peptic ulcer disease, inflammatory bowel disease, or other gastrointestinal condition increasing the risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to beginning therapy.
* Presence of uncontrolled infection.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib.
* Corrected QT interval (QTc) prolongation defined as QTc interval > 470 msecs.
* History of any one of the following cardiac conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* History of cerebrovascular accident or pulmonary embolus within the past 6 months.
* Has Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system (See Appendix 6)
* Poorly controlled hypertension (systolic blood pressure (SBP) of ≥ 140mmHg, or diastolic blood pressure (DBP) of ≥ 90mmHg).
* Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. The blood pressure (BP) must be re-assessed on two occasions that are separated by a minimum of 24 hours. The mean SBP/DBP values from both BP assessments must be < 140/90mmHg in order for a subject to be eligible for the study.
* History of untreated deep venous thrombosis (DVT) within the past 6 months (e.g. calf vein thrombosis).
* Note: Patients with recent DVT who are treated with therapeutic anti-coagulant agents (excluding therapeutic warfarin) for at least 6 weeks are eligible.
* Presence of any non-healing, non-tumor related wound, fracture, or ulcer, or the presence of symptomatic peripheral vascular disease.
* Subjects with bilateral hydronephrosis which cannot be alleviated by ureteral stents or percutaneous drainage.
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to beginning therapy, or anticipation of the need for a major surgical procedure during the course of the study; minor surgical procedures such as fine needle aspiration or core biopsy within 1 week prior to beginning therapy are also excluded.
* Unable to swallow and retain orally administered medication.
* Pregnant or lactating female.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (60):
- United States (12):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Dallas, Texas
- Argentina (7):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Neuquén, Neuquén Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santa Fe, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Quilmes
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Canada (5):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (6):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Villejuif
- Germany (5):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Saarbrücken, Saarland
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
- India (4):
  - GSK Investigational Site, Ahemdabad
  - GSK Investigational Site, Mangalore
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Trivandrum
- Ireland (2):
  - GSK Investigational Site, Cork
  - GSK Investigational Site, Dublin
- Italy (4):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Campobasso, Molise
- GSK Investigational Site, Mexico City, Mexico
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, La Laguna (Santa Cruz de Tenerife)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Pamplona
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen

REFERENCES:
- [Result] Monk BJ, Mas Lopez L, Zarba JJ, Oaknin A, Tarpin C, Termrungruanglert W, Alber JA, Ding J, Stutts MW, Pandite LN. Phase II, open-label study of pazopanib or lapatinib monotherapy compared with pazopanib plus lapatinib combination therapy in patients with advanced and recurrent cervical cancer. J Clin Oncol. 2010 Aug 1;28(22):3562-9. doi: 10.1200/JCO.2009.26.9571. Epub 2010 Jul 6. PMID 20606083
- [Result] Monk BJ, Pandite LN. Survival data from a phase II, open-label study of pazopanib or lapatinib monotherapy in patients with advanced and recurrent cervical cancer. J Clin Oncol. 2011 Dec 20;29(36):4845. doi: 10.1200/JCO.2011.38.8777. Epub 2011 Nov 14. No abstract available. PMID 22084371
- [Derived] de Jonge MJ, Hamberg P, Verweij J, Savage S, Suttle AB, Hodge J, Arumugham T, Pandite LN, Hurwitz HI. Phase I and pharmacokinetic study of pazopanib and lapatinib combination therapy in patients with advanced solid tumors. Invest New Drugs. 2013 Jun;31(3):751-9. doi: 10.1007/s10637-012-9885-8. Epub 2012 Oct 6. PMID 23054212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) continued to be enrolled into all three treatment arms after clinical data cutoff for the interim analysis, but before the results were evaluated. Final total enrollment was 228 participants: 76 in the combination arm, 78 in the lapatinib monotherapy arm, and 74 in the pazopanib monotherapy arm.
Pre-assignment Details: Study was initially designed and started as a randomized, three-arm, controlled trial. Participants were randomized to the combination of pazopanib plus lapatinib, pazopanib monotherapy, or lapatinib monotherapy. Based on results from a planned interim analysis, the combination group was terminated, but the monotherapy groups continued as planned.
Groups:
- Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg: Lapatinib 1500 mg (6 x 250 mg tablets) and pazopanib 800 mg (2 x 400 mg tablets) daily
- Lapatinib Monotherapy: 1500 mg (6 x 250 mg tablets) of oral lapatinib daily
- Pazopanib Monotherapy: 800 mg (2 x 400 mg tablets) of oral pazopanib daily
Period: Interim Analysis; 11 February 2008
Arm/Group | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg | Lapatinib Monotherapy | Pazopanib Monotherapy
Started | 59 | 58 | 60
Ongoing | 23 | 20 | 25
Completed | 0 | 0 | 0
Not Completed | 59 | 58 | 60
Not completed — Adverse Event | 10 | 3 | 7
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 2
Not completed — Sponsor Terminated Study | 1 | 0 | 0
Not completed — Disease Progression | 16 | 30 | 22
Not completed — Death | 0 | 1 | 0
Not completed — Par. Withdrew; Followed for Survival | 2 | 0 | 0
Not completed — Physician Decision | 2 | 3 | 3
Not completed — Ongoing | 23 | 20 | 25
Period: Final Analysis; 31 July 2008
Arm/Group | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg | Lapatinib Monotherapy | Pazopanib Monotherapy
Started | 0 | 78 | 74
Ongoing | 0 | 29 | 32
Completed | 0 | 39 | 26
Not Completed | 0 | 39 | 48
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 7
Not completed — Physician Decision | 0 | 6 | 6
Not completed — Other | 0 | 1 | 0
Not completed — Ongoing | 0 | 29 | 32
Period: End-of-Study Analysis; 28 July 2011
Arm/Group | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg | Lapatinib Monotherapy | Pazopanib Monotherapy
Started | 77 (Enrollment continued in this arm after data cut for Interim Analysis and before arm closed.) | 77 (1 participant randomized to lapatinib (final analysis table) actually received combination therapy.) | 74
Completed | 53 | 59 | 54
Not Completed | 24 | 18 | 20
Not completed — Lost to Follow-up | 5 | 3 | 3
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 7
Not completed — Sponsor Terminated Study | 4 | 5 | 4
Not completed — Physician Decision | 4 | 6 | 6
Not completed — Other | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg | Lapatinib Monotherapy | Pazopanib Monotherapy | Total
Number analyzed (Participants) | 59 | 58 | 60 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Interim Analysis
  years | 50.4 (11.04) | 48.7 (11.47) | 49.6 (10.34) | 49.5 (10.91)
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Final Analysis (n=0, 78, 74)
  years | NA (NA) — There are no participants for this analysis subgroup. | 49.2 (11.27) | 50.8 (10.93) | 50 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at Interim Analysis
  Participants
    Female | 59 | 58 | 60 | 177
    Male | 0 | 0 | 0 | 0
Gender [Number; unit: participants] — Gender at Final Analysis (n=0, 78, 74)
  participants
    Female | NA — There are no participants for this analysis subgroup. | 78 | 74 | 152
    Male | NA — There are no participants for this analysis subgroup. | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Race at Interim Analysis
  participants
    African American | 0 | 1 | 0 | 1
    American Indian | 10 | 4 | 12 | 26
    Asian-South East | 12 | 10 | 8 | 30
    White | 37 | 43 | 40 | 120
Race/Ethnicity, Customized [Number; unit: participants] — Race at Final Analysis (n=0, 78, 74)
  participants
    African American | NA — There are no participants for this analysis subgroup. | 1 | 0 | 1
    American Indian | NA — There are no participants for this analysis subgroup. | 10 | 13 | 23
    Asian-Central , South | NA — There are no participants for this analysis subgroup. | 2 | 0 | 2
    Asian-South East | NA — There are no participants for this analysis subgroup. | 13 | 9 | 22
    White | NA — There are no participants for this analysis subgroup. | 52 | 52 | 104
Histology at diagnosis: Interim Analysis [Number; unit: participants]
  Adenocarcinoma | 15 | 8 | 8 | 31
  Adenosquamous carcinoma | 0 | 4 | 3 | 7
  Squamous cell carcinoma | 32 | 38 | 43 | 113
  Other | 10 | 8 | 5 | 23
  Missing | 2 | 0 | 1 | 3
Histology at diagnosis: Final Anaysis [Number; unit: participants] — (n=0, 78, 74)
  participants
    Adenocarcinoma | NA — There are no participants for this analysis subgroup. | 11 | 12 | 23
    Adenosquamous carcinoma | NA — There are no participants for this analysis subgroup. | 4 | 3 | 7
    Squamous cell carcinoma | NA — There are no participants for this analysis subgroup. | 55 | 53 | 108
    Other | NA — There are no participants for this analysis subgroup. | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) in Interim Analysis
Description: PFS is defined as the interval between the date of randomization and the date of disease progression or death due to any cause. The study was designed to test Combination vs. Lapatinib first. The result indicated that Combination would not show improvement over Lapatinib even if followed until the final analysis and the Combination arm was terminated. The monotherapy arms continued to the final analysis. Data shown here are from this interim analysis.
Time Frame: From randomization until at least 35 PFS events in pairwise comparison of the three treatment arms (Interim Analysis; up to 52.14 weeks)
Population: Intent to Treat (ITT) Population: all randomized participants
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg | Lapatinib Monotherapy | Pazopanib Monotherapy
Number analyzed (Participants) | 59 | 58 | 60
Weeks | 12.6 [11.7 to 14.1] | 12.6 [11.6 to 18.3] | 17.9 [12.1 to 23.9]
Statistical Analysis 1: Comparison: Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg vs Lapatinib Monotherapy; Test type: Superiority or Other; p = 0.535, Log Rank — Stratified log-rank test with one-sided p-value. p<=0.0037 required for significance, and p>0.4956 indicated futility; Hazard Ratio (HR) = 1.05, 90% CI [0.65 to 1.7] — The estimated value is the hazard ratio comparing combination to lapatinib monotherapy

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization until death due to any cause.
Time Frame: From Randomization (11 December 2006) until approximately 78% overall survival events at the time of the second overall survival update (3 March 2010) (up to 168.29 weeks)
Population: ITT Population
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Lapatinib Monotherapy | Pazopanib Monotherapy
Number analyzed (Participants) | 78 | 74
Weeks | 44.1 [35.6 to 48.9] | 49.7 [42.0 to 55.9]

3. Secondary Outcome: Clinical Benefit Response
Description: Clinical benefit response is defined as the number of participants with evidence of complete (CR) or partial (PR) tumor response or stable disease (SD) for at least 6 months (183 days). Per Response Evaluation Criteria In Solid Tumors (RECIST): CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum; Stable Disease, small changes that do not meet previously given criteria. Confirmation requires at least 2 assessments of CR/PR with at least 4 weeks between assessments.
Time Frame: From Randomization until 105 total PFS events in combined population of two monotherapy arms (up to 85.57 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib Monotherapy | Pazopanib Monotherapy
Number analyzed (Participants) | 78 | 74
participants | 7 | 15

4. Secondary Outcome: Response
Description: Response is defined as the number of participants achieving either a complete or partial tumor response per RECIST criteria. CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum.
Time Frame: From Randomization until 105 total PFS events in combined population of two monotherapy arms (up to 85.57 weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib Monotherapy | Pazopanib Monotherapy
Number analyzed (Participants) | 78 | 74
participants | 4 | 7
Statistical Analysis 1: Comparison: Lapatinib Monotherapy vs Pazopanib Monotherapy; Test type: Superiority or Other; p = 0.237, Fisher Exact — One-sided p-value

5. Secondary Outcome: Time to Response
Description: For the subset of participants who showed a confirmed CR or PR, time to response was defined as the time from randomization until the first documented evidence of CR or PR (whichever status was recorded first). CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum.
Time Frame: From Randomization until 105 total PFS events in combined population of two monotherapy arms (up to 85.57 weeks)
Population: ITT Population
Measure: Mean (90% Confidence Interval); unit: weeks
Arm/Group | Lapatinib Monotherapy | Pazopanib Monotherapy
Number analyzed (Participants) | 4 | 7
weeks | 18.2 [6.0 to 24.1] | 6.9 [5.6 to 11.9]

6. Secondary Outcome: Duration of Response
Description: For participants who had a CR or PR, the duration of response was defined as the time from first documented evidence of PR or CR until the first documented sign of disease progression or death. CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum.
Time Frame: From Randomization until 105 total PFS events in combined population of two monotherapy arms (up to 85.57 weeks)
Population: ITT Population. The median for lapatinib was not reached at the time of data cut-off. No formal analysis of this endpoint was conducted for this group due to a very small number of responding participants.
Measure: Mean (90% Confidence Interval); unit: weeks
Arm/Group | Lapatinib Monotherapy | Pazopanib Monotherapy
Number analyzed (Participants) | 0 | 7
weeks |  | 48.1 [12.0 to 48.1]

7. Secondary Outcome: Safety and Tolerability of Pazopanib, Lapatinib and the Combination of Pazopanib and Lapatinib
Description: Safety was assessed as the number of participants experiencing a serious adverse event (SAE) or an adverse event (AE). See the adverse event module for safety data.
Time Frame: From Randomization (11 December 2006) until last participant had last visit (28 July 2011) in combined population of two monotherapy arms (up to 241.43 weeks)
Population: Safety Population: all participants who received at least one dose of study drug
Measure: Number; unit: participants
Groups:
- Combination Therapy: Lapatinib 1500 mg and Pazopanib 800: Lapatinib 1500 mg (6 x 250 mg tablets) and pazopanib 800 mg (2 x 400 mg tablets) daily
Arm/Group | Lapatinib Monotherapy | Pazopanib Monotherapy | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800
Number analyzed (Participants) | 76 | 74 | 76
participants
  Serious adverse events | 22 | 28 | 32
  Other adverse events with >5% occurrence | 66 | 69 | 71

8. Primary Outcome: Progression-free Survival (PFS) in Final Analysis
Description: PFS is defined as the interval between the date of randomization and the date of disease progression or death due to any cause. This study began as a 3-arm study. The combination arm was terminated at the interim analysis. The monotherapy arms continued to final analysis. Data shown here are from the final analysis.
Time Frame: From Randomization until 105 total PFS events in combined population of two monotherapy arms (up to 85.57 weeks)
Population: ITT Population
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Lapatinib Monotherapy | Pazopanib Monotherapy
Number analyzed (Participants) | 78 | 74
Weeks | 17.1 [12.1 to 18.1] | 18.1 [15.1 to 24.6]
Statistical Analysis 1: Comparison: Lapatinib Monotherapy vs Pazopanib Monotherapy; Test type: Superiority or Other; p = 0.013, Log Rank — Stratified log-rank test with one-sided p-value; Hazard Ratio, log = 0.66, 90% CI [0.48 to 0.91]

ADVERSE EVENTS:
Time Frame: SAEs/AEs were assessed in par. receiving >=1 dose of study treatment at time of final PFS analysis (From Randomization [11 December 2006] until last par. had last visit [28 July 2011] in combined population of two monotherapy arms [up to 241.43 weeks])
Description: Serious adverse events (SAEs) and adverse events (AEs) are reported for the Safety Population (all participants who received at least one dose of study drug).
Arm/Group | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg | Lapatinib Monotherapy | Pazopanib Monotherapy
Serious Adverse Events (participants affected / at risk) | 32/76 | 22/76 | 28/74
Other Adverse Events (participants affected / at risk) | 71/76 | 66/76 | 69/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg (N=76) | Lapatinib Monotherapy (N=76) | Pazopanib Monotherapy (N=74)
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 4
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Pyonephrosis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 4 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 1
Cervix disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Chest pain (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Performance status decreased (General disorders) | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 2
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0 | 0
Urethral fistula (Renal and urinary disorders) | 1 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Genital hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Lapatinib 1500 mg and Pazopanib 800 mg (N=76) | Lapatinib Monotherapy (N=76) | Pazopanib Monotherapy (N=74)
Diarrhoea (Gastrointestinal disorders) | 58 | 42 | 40
Nausea (Gastrointestinal disorders) | 28 | 25 | 28
Vomiting (Gastrointestinal disorders) | 32 | 18 | 15
Abdominal pain (Gastrointestinal disorders) | 15 | 9 | 14
Constipation (Gastrointestinal disorders) | 8 | 8 | 17
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7 | 13
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 4 | 5 | 2
Asthenia (General disorders) | 19 | 17 | 13
Fatigue (General disorders) | 14 | 15 | 10
Oedema peripheral (General disorders) | 5 | 8 | 6
Pain (General disorders) | 3 | 1 | 5
Pyrexia (General disorders) | 5 | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 12 | 22 | 4
Hair colour changes (Skin and subcutaneous tissue disorders) | 8 | 0 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 5 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 1 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 5
Acne (Skin and subcutaneous tissue disorders) | 6 | 4 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 4 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 11 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 7 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 29 | 25 | 20
Urinary tract infection (Infections and infestations) | 9 | 10 | 6
Pharyngitis (Infections and infestations) | 0 | 0 | 4
Headache (Nervous system disorders) | 10 | 7 | 20
Dizziness (Nervous system disorders) | 3 | 5 | 5
Dysgeusia (Nervous system disorders) | 11 | 3 | 5
Blood alkaline phosphatase increased (Investigations) | 7 | 5 | 14
Aspartate aminotransferase increased (Investigations) | 9 | 2 | 11
Alanine aminotransferase increased (Investigations) | 5 | 1 | 11
Blood lactate dehydrogenase increased (Investigations) | 5 | 1 | 8
Weight decreased (Investigations) | 6 | 4 | 3
Hypertension (Vascular disorders) | 24 | 2 | 23
Anaemia (Blood and lymphatic system disorders) | 12 | 12 | 8
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 9
Leukopenia (Blood and lymphatic system disorders) | 6 | 0 | 5
Proteinuria (Renal and urinary disorders) | 9 | 11 | 6
Dysuria (Renal and urinary disorders) | 5 | 4 | 3
Haematuria (Renal and urinary disorders) | 3 | 5 | 3
Pelvic pain (Reproductive system and breast disorders) | 4 | 5 | 5
Vaginal haemorrhage (Reproductive system and breast disorders) | 8 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2
Insomnia (Psychiatric disorders) | 3 | 5 | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 4 | 2
Flatulence (Gastrointestinal disorders) | 1 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 8 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 5 | 1
Somnolence (Nervous system disorders) | 0 | 4 | 3
Haemoglobin decreased (Investigations) | 2 | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 4
Urinary incontinence (Renal and urinary disorders) | 0 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.